CLINICAL TRIAL: NCT06756815
Title: Effects of Cross Bracing Protocol With And Without Dynamic Neuromuscular Stabilization Training on Functional Movements in Athletes With Acute Anterior Cruciate Ligament Injury
Brief Title: Cross Bracing Protocol With And Without Dynamic Neuromuscular Stabilization Training in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0420
Record Dates: First submitted 2024-11-18; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Sports Physical Therapy
Keywords: Anterior Cruciate Ligament; cross brace movement; dynamic stabilization; Functional movement
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Cross bracing + conservative treatment(control group) (Experimental): Cross brace training week 1-2 1. Cross Bracing (Isometric Holds) 2. Quad Sets 3. Straight Leg Raise 4. Ankle Pumps 5. Heel and Toe Raises 6. Glute Bridge Week 3-4
  1. Cross Bracing (Isometric Holds)
  2. Hamstring Curls
  3. Step-ups
  4. Mini Squats (with support)
  5. Leg Press
  6. Lateral Leg Raises Week 5-6
  1. Cross Bracing (Isometric Holds) 2. Single-leg Balance (with support) 3. Lunges (with proper technique) 4. Squats (bodyweight) 5. Box Jumps 6. Lateral Step-ups
  Interventions: Other: Cross bracing and conservative treatment
- Group B: Cross bracing + DNS training + conservative treatment (Experimental): Week 1-2
  1. Cross Bracing (Isometric Holds)
  2. DNS Core Activation (supine, prone positions)
  3. Quad Sets
  4. Straight Leg Raise
  5. Ankle Pumps
  6. Heel and Toe Raises
  7. Glute Bridge Week 3-4
  1. Cross Bracing (Isometric Holds) 2. DNS Core Stabilization (advanced activation) 3. Hamstring Curls 4. Step-ups 5. Mini Squats 6. Leg Press 7. Lateral Leg Raises 8. Pelvic Tilts Week 5-6
  1. Cross Bracing (Isometric Holds)
  2. DNS Dynamic Stabilization (with resistance)
  3. Single-leg Balance (with and without support)
  4. Lunges (with added resistance)
  5. Squats (bodyweight or weighted)
  6. Box Jumps
  7. Lateral Step-ups
  8. Running Drills (if tolerated)
  Interventions: Other: Cross bracing and DNS with conservative treatment

INTERVENTIONS:
Other: Cross bracing and conservative treatment — Week Exercise Training Frequency (sets x reps) Week 1-2 1. Cross Bracing (Isometric Holds) 2. Quad Sets 3. Straight Leg Raise 4. Ankle Pumps 5. Heel and Toe Raises 6. Glute Bridge 2 sets x 10 reps Week 3-4 1. Cross Bracing (Isometric Holds) 2. Hamstring Curls 3. Step-ups 4. Mini Squats (with support) 5. Leg Press 6. Lateral Leg Raises 3 sets x 12 reps Week 5-6 1. Cross Bracing (Isometric Holds) 2. Single-leg Balance (with support) 3. Lunges (with proper technique) 4. Squats (bodyweight) 5. Box Jumps 6. Lateral Step-ups 3 sets x 15 reps
  Other Names: • Landing Error Scoring System; • International Knee Documentation Committee (IKDC) score; • Functional Movement Screening
  Arms: Group A: Cross bracing + conservative treatment(control group)
Other: Cross bracing and DNS with conservative treatment — Week Exercise Training Frequency (sets x reps) Week 1-2
  1. Cross Bracing (Isometric Holds)
  2. DNS Core Activation (supine, prone positions)
  3. Quad Sets
  4. Straight Leg Raise
  5. Ankle Pumps
  6. Heel and Toe Raises
  7. Glute Bridge 2 sets x 10 reps Week 3-4
  1. Cross Bracing (Isometric Holds) 2. DNS Core Stabilization (advanced activation) 3. Hamstring Curls 4. Step-ups 5. Mini Squats 6. Leg Press 7. Lateral Leg Raises 8. Pelvic Tilts 3 sets x 12 reps Week 5-6
  1. Cross Bracing (Isometric Holds)
  2. DNS Dynamic Stabilization (with resistance)
  3. Single-leg Balance (with and without support)
  4. Lunges (with added resistance)
  5. Squats (bodyweight or weighted)
  6. Box Jumps
  7. Lateral Step-ups
  8. Running Drills (if tolerated) 3 sets x 15 reps
  Arms: Group B: Cross bracing + DNS training + conservative treatment

SUMMARY:
ACL Injury is a severe injury for athletes, which frequently results in functional limits and a higher likelihood of re-injury. Although bracing regimens are frequently used in rehabilitation, their ability to restore functional movements after an ACL Injury is still uncertain. Dynamic neuromuscular stabilization (DNS) training, which targets the core and proprioception, has emerged as a viable method for enhancing motor control and decreasing knee instability. The objective of this study is to examine the synergistic impact of cross bracing and DNS training on the functional movements of athletes who have recently experienced an ACL Injury .

A randomized controlled trial will be conducted to study the effects of different interventions on athletes with acute ACL Injury. The participants will be divided into two groups: (A= control group) Cross bracing with conservative treatment, (B= Treatment group) Cross bracing + DNS training with conservative treatment. Both groups will engage in targeted exercises that aim to activate the core, improve proprioception, and enhance movement patterns. The participants' functional movements will be assessed at the beginning of the study and 6 weeks later using established questionnaire such as International Knee Documentation Committee (IKDC) score - assesses knee function and symptoms, Landing error scoring system (LESS), Y Balance (YB), Functional movement screening (FMS) Statistical analysis will be performed to compare the functional performance and neuromuscular parameters between the groups in order to determine the most effective intervention for restoring movement quality after ACL Injury .

DETAILED DESCRIPTION:
The study's emphasis on cross bracing protocol and DNS training is warranted due to the necessity of investigating non-invasive and conservative therapy methods that have the ability to improve functional movements in athletes with ACL Injury . Cross bracing is frequently employed to offer external reinforcement and enhance stability to the knee joint subsequent to an ACL damage, whereas DNS training concentrates on reconditioning the neuromuscular system to enhance movement patterns and motor control. The study seeks to provide significant insights into the most effective rehabilitation regimens for athletes with acute ACL Injury by evaluating the effects of two therapies. The ultimate goal is to enhance their functional results and long-term sports performance.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* Age: 18-30 years.
* Mentally and verbally capable of participating in the study.
* Positive Lachman Test
* Diagnosis of acute ACL Injury with grade 1 and 2 through MRI or arthroscopy.

Exclusion Criteria:

* Inflammatory disease, rheumatoid arthritis, spondyloarthropathy or active malignancy.
* Neurological disorder or systemic disease.
* Previous surgery on the affected knee.
* Meniscal tear or articular cartilage damage requiring surgical repair

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
International Knee Documentation Committee score | 6 week
  The International Knee Documentation Committee (IKDC) Subjective Knee Form is a patient-oriented questionnaire that assesses symptoms and function in daily living activities. The purpose of this study was to validate the IKDC Subjective Knee Form in a large patient population with various knee disorders. It contains sections on knee symptoms (7 items), function (2 items), and sports activities (2 items). Scores range from 0 points (lowest level of function or highest level of symptoms) to 100 points (highest level of function and lowest level of symptoms). The overall IKDC score showed acceptable test-retest reliability with an interclass correlation of 0.95.
Landing Error Scoring System | 6 week
  The Landing Error Scoring System (LESS) is a clinical tool often used in research and practice to identify athletes presenting high injury-risk biomechanical patterns during a jump-landing task. It is used to identify the risk of non-contact injuries during jumping and landing movements. It assesses 9 landing concepts and has 17 questions which are scored out of 19 points. Interrater reliability (ICC2, 1) for the LESS-RT ranged from .72 to .81 with standard error of measurements ranging from .69 to .79.
Y- Balance Test | 6 week
  The Y Balance Test was developed as a test of dynamic postural control and has been shown to be predictive of lower-extremity injury. It can be used for both the upper quarter and lower quarter. The YBT for the lower quarter (LQYBT) has been thoroughly researched as its protocol is based on research done on the Star Excursion Balance Test. The Star Excursion Balance Test demonstrated reliable results on its ability to predict LE injury in high school basketball players. The YBT has proven to have very good levels of interrater test-retest reliability (ICC = 0.80 - 0.85)
Functional Movement Screening | 6 week
  The Functional Movement Screen (FMS) is utilized by professional and collegiate sports teams and the military for the prevention of musculoskeletal injuries. The FMS is a tool used to identify asymmetries which result in functional movement deficiencies. The FMS aims to identify imbalances in mobility and stability during seven fundamental movement patterns. ICC values of 0.90-0.99 indicated excellent reliability, 0.80-0.89 indicated good reliability, 0.70-0.79 indicated fair reliability, and 0-0.69 indicated poor reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- PSRD, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang XG, Feng JT, He X, Wang F, Hu YC. The effect of knee bracing on the knee function and stability following anterior cruciate ligament reconstruction: A systematic review and meta-analysis of randomized controlled trials. Orthop Traumatol Surg Res. 2019 Oct;105(6):1107-1114. doi: 10.1016/j.otsr.2019.04.015. Epub 2019 Jul 3. PMID 31279767
- [Background] Mahdieh L, Zolaktaf V, Karimi MT. Effects of dynamic neuromuscular stabilization (DNS) training on functional movements. Hum Mov Sci. 2020 Apr;70:102568. doi: 10.1016/j.humov.2019.102568. Epub 2020 Jan 13. PMID 31950895
- [Background] Raines BT, Naclerio E, Sherman SL. Management of Anterior Cruciate Ligament Injury: What's In and What's Out? Indian J Orthop. 2017 Sep-Oct;51(5):563-575. doi: 10.4103/ortho.IJOrtho_245_17. PMID 28966380
- [Background] Filbay SR, Grindem H. Evidence-based recommendations for the management of anterior cruciate ligament (ACL) rupture. Best Pract Res Clin Rheumatol. 2019 Feb;33(1):33-47. doi: 10.1016/j.berh.2019.01.018. Epub 2019 Feb 21. PMID 31431274
- [Background] Dunphy E, Button K, Hamilton F, Williams J, Spasic I, Murray E. Feasibility randomised controlled trial comparing TRAK-ACL digital rehabilitation intervention plus treatment as usual versus treatment as usual for patients following anterior cruciate ligament reconstruction. BMJ Open Sport Exerc Med. 2021 May 5;7(2):e001002. doi: 10.1136/bmjsem-2020-001002. eCollection 2021. PMID 34035951
- [Background] Greenberg EM, Greenberg ET, Albaugh J, Storey E, Ganley TJ. Anterior Cruciate Ligament Reconstruction Rehabilitation Clinical Practice Patterns: A Survey of the PRiSM Society. Orthop J Sports Med. 2019 Apr 23;7(4):2325967119839041. doi: 10.1177/2325967119839041. eCollection 2019 Apr. PMID 31041331
- [Background] Book E, Noyes FR, editors. Read Online The Anterior Cruciate Ligament Reconstruction And Basic Science E Book Anterior Cruciate Ligament: Reconstruction and Basic Science2022.
- [Background] Filbay SR, Dowsett M, Chaker Jomaa M, Rooney J, Sabharwal R, Lucas P, Van Den Heever A, Kazaglis J, Merlino J, Moran M, Allwright M, Kuah DEK, Durie R, Roger G, Cross M, Cross T. Healing of acute anterior cruciate ligament rupture on MRI and outcomes following non-surgical management with the Cross Bracing Protocol. Br J Sports Med. 2023 Dec;57(23):1490-1497. doi: 10.1136/bjsports-2023-106931. Epub 2023 Jun 14. PMID 37316199
- [Background] Karimijashni M, Sarvestani FK, Yoosefinejad AK. The Effect of Contralateral Knee Neuromuscular Exercises on Static and Dynamic Balance, Knee Function, and Pain in Athletes Who Underwent Anterior Cruciate Ligament Reconstruction: A Single-Blind Randomized Controlled Trial. J Sport Rehabil. 2023 Mar 14;32(5):524-539. doi: 10.1123/jsr.2021-0380. Print 2023 Jul 1. PMID 36918020